CLINICAL TRIAL: NCT06606496
Title: Comparison of the Effect of Testosterone Administered for Micropenis Hypospadias Surgery With Bispectral Index and Other Parameters in General Anesthesia: A Prospective Observational Study
Brief Title: Comparison of the Effect of Testosterone Administered for Micropenis Hypospadias Surgery With Bispectral Index
Status: Not yet recruiting | Type: Observational
Sponsor: Namik Kemal University (Other)
Responsible Party: Principal Investigator, Ahmet Gültekin, Associate Professor, Namik Kemal University
Other Study IDs: NamikKU-AGultekin-1
Record Dates: First submitted 2024-09-13; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: General Anesthesia; Testosterone; BIS
MeSH Terms: interventions — Consciousness Monitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Group Control (Group K)
- Group Testosterone (Group T)
  Interventions: Device: Bispectral index (BIS)

INTERVENTIONS:
Device: Bispectral index (BIS) — The bispectral index (BIS) monitor is a quantitative electroencephalographic (EEG) device that is widely used to assess the hypnotic component of anaesthesia, especially when neuromuscular blocking drugs are used. If necessary, it may be necessary to increase or decrease MAC (minimum alveolar concentration) in the testosterone group according to the BIS monitoring value.
  Groups: Group Testosterone (Group T)

SUMMARY:
The aim of this observational study is to learn the effects of hormone therapy (testosterone) applied in micropenis hypospadias surgery on the depth of anesthesia under general anesthesia. The main question it aims to answer is: The effect of testosterone therapy on the depth of general anesthesia. Based on these, to comment on the depth of anesthesia of patients who have just started using testosterone for sex change. To follow the depth of anesthesia of patients who have undergone hypospadias surgery with BIS monitoring and to record respiratory parameters under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Ages 1-16
* Patients with ASA I (Normal healthy patients except for surgery)
* Patients who will undergo surgery for hypospadias repair

Exclusion Criteria:

* Morbidly obese patients (body mass index > 40kg/m2)
* ASA II-III-IV patients (other groups of patients with additional diseases)
* Volunteers who do not want to participate in the study

Ages: 1 Year to 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients undergoing hypospadias repair surgery
Sampling Method: Probability Sample
Enrollment: 22 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
BIS values | 4 months
  in addition to monitoring the MAC and vital values in order to monitor the depth of anesthesia, BIS monitoring values, which are a special EEG parameter and can be continuously monitored throughout the surgery, also provide better quality results. The use of the BIS monitor reduces the incidence of awareness under anesthesia. The fact that the procedure is non-invasive is an advantage in terms of use.
  Hypospadias often requires surgical intervention. Before this surgical intervention, pediatric surgeons perform hormone (testosterone) treatment (IM) in patients with micropenis to temporarily enlarge the penis size, which affects the success of the surgery. It is usually applied intramuscularly one week before the surgery in a pediatric surgery clinic.
  Some studies have reported that anesthetic requirements change with testosterone changes (to provide sufficient depth of anesthesia with changes in the depth of anesthesia).

SECONDARY OUTCOMES:
sex change and anesthesia | 4 months
  Comment on the initial anesthesia of adult patients who have to use testosterone after sex change